CLINICAL TRIAL: NCT07356232
Title: Partial Enteral Nutrition as Therapeutic Augmentation of Advanced Pharmacological Therapy in Patients With Active Crohn's Disease
Acronym: PANDORA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 859860
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease, Active
Keywords: partial enteral nutrition; Crohn's disease exclusion diet
MeSH Terms: conditions — Crohn Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial enteral nutrition (Experimental): Participants will consume Kate Farms Peptide 1.5 for 60% of their calories for 8 weeks
  Interventions: Dietary Supplement: Partial enteral nutrition - orally consumed formula
- No partial enteral nutrition (No Intervention)

INTERVENTIONS:
Dietary Supplement: Partial enteral nutrition - orally consumed formula — Participants will consume Kate Farms Peptide 1.5 for approximately 60% of their calories while following the Crohn's Disease Exclusion Diet.
  Arms: Partial enteral nutrition

SUMMARY:
This is a multicenter non-randomized prospective open label trial of partial enteral nutrition (PEN) among patients with active Crohn's disease (CD) starting standard of care advanced therapy. Our central hypothesis is that combination therapy of PEN and pharmacologic therapy is more efficacious than pharmacologic therapy alone and can be well-tolerated for patients. Participants will choose to either include PEN along with starting their advanced therapy or will choose not to include PEN. 80 participants will be recruited from 15 sites across the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. A confirmed diagnosis of Crohn's disease
3. Plan to start one advanced Crohn's Disease therapy (anti-TNF, anti-IL12/IL23, anti-IL23, anti-alpha 4 beta 7, JAK inhibitor). Methotrexate, aminosalicylates and thiopurines are permitted to be continued with the advanced therapy if on stable dose for at least 8 weeks. Methotrexate or thiopurines may be initiated within 1 week of starting the advanced pharmacologic therapy.
4. Active disease defined by at least one of the criteria from group A AND one from group B.

Group A

1. Short Crohn's Disease Activity Index (sCDAI) score >1758
2. sCDAI < 175 and on 10- 30 mg of prednisone (or 6-9 mg of budesonide) at a stable dose for 2 weeks. Stable daily dose of corticosteroids cannot exceed prednisone 30 mg or budesonide 9 mg. Must have experienced worsening of symptoms with attempts to taper to a lower dose of steroids in 3 months prior to screening.

Group B

1. Fecal calprotectin at baseline ≥ 300 ug/gr
2. Active disease seen at colonoscopy within 8 weeks of the screening visit. Active disease requires presence of mucosal breaks including either diffuse scattered erosions or at least one ulcer (>5mm diameter)
3. Active disease on cross-sectional imaging (CT scan, MRI or ultrasound) within 8 weeks of the screening visit (evidence of acute inflammation, such as ulceration or bowel wall thickening with restricted diffusion)

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Presence of an ostomy
3. Previous total colectomy
4. Short gut syndrome from prior surgeries
5. Consuming parenteral nutrition for more than 350 calories per day in the two weeks prior to screening
6. Having been on the Crohn's Disease Exclusion Diet (CDED) in the 2 weeks prior to screening
7. Plan to receive two simultaneously administered advanced therapies
8. Planning to start a new medication in the same class as the medication currently taking. This does not include a switch from Ustekinumab to anti-IL23 drugs.
9. Impending need for CD surgery per investigator
10. Symptomatic stricture or stricture inducing bowel dilation as per local investigator.
11. >4 very soft or liquid bowel movements per day when feeling well
12. Diabetes mellitus requiring therapy with medication
13. Known allergy to any ingredient in the Kate Farms formula.
14. Previous therapy with EEN or PEN for a minimum of two consecutive weeks- defined as over 60% of calories from PEN
15. Unable to receive shipments of PEN formula.
16. Starting a new medication for Crohn's disease other than steroids in the 8 weeks prior to the screening visit
17. Starting an accelerated (non-FDA approved) dose of advanced therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Rate of steroid-free remission following 8 weeks of pharmacologic therapy | From start of pharmacologic therapy to 8 weeks.
  Steroid-free clinical remission at Visit 5 (week 8) of pharmacologic therapy initiation will be defined as a short Crohn's Disease Activity Index (sCDAI) < 150 points while off steroids. The need to switch therapies, increase or initiate corticosteroids or any other CD drug will be considered as a failure to achieve the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No